CLINICAL TRIAL: NCT01422473
Title: Hemorrhoidectomy Using the Enseal Device: A Comparison to Open Hemorrhoidectomy Techniques
Brief Title: Comparison Study of Hemorrhoid Surgery Using the Enseal Device to Standard Hemorrhoid Surgical Techniques
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Terminated due to poor accrual.
Sponsor: Swedish Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IR 4957
Record Dates: First submitted 2011-08-22; First posted 2011-08-24 (Estimated); Last update posted 2013-06-05 (Estimated); Status verified 2013-06

CONDITIONS: Hemorrhoids
Keywords: Hemorrhoids; Rectal Diseases; Intestinal Diseases; Gastrointestinal Diseases; Digestive System Diseases
MeSH Terms: conditions — Hemorrhoids; Rectal Diseases; Intestinal Diseases; Gastrointestinal Diseases; Digestive System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- EnSeal Device (Experimental): EnSeal Trio Tissue Sealing Device
  Interventions: Device: EnSeal Trio Tissue Sealing Device

INTERVENTIONS:
Device: EnSeal Trio Tissue Sealing Device — For surgery in ligating and dividing vascular tissue during abdominal surgery.

SUMMARY:
The purpose of this study is to examine the advantages and disadvantages of using the EnSeal device in hemorrhoid surgery as compared to traditional hemorrhoid surgery techniques.

It is hypothesized that the use of the Enseal device will demonstrate an improvement a patient's overall experience through less postoperative bleeding and pain, decreased time for wound healing, and a faster return to work.

DETAILED DESCRIPTION:
The EnSeal Device is FDA approved for surgery in ligating and dividing vascular tissue during abdominal surgery. Electrical energy is converted into heat energy and resultant simultaneous division of tissues. This allows surgery to be bloodless and sutureless. It has been successfully used by many individual practitioners for hemorrhoidectomy, with apparent advantage and success; but to date, no comparative study has been done to assess the advantages and disadvantages of this method of hemorrhoidectomy, when compared to traditional excisional techniques. The investigators propose to use this device in the current study in the treatment of hemorrhoidal disease where vascular tissue is excised in bloodless and sutureless fashion. It is currently being used in institutions throughout the United States and Europe.

After surgery, patients will receive the same standard postoperative instructions as for conventional hemorrhoidectomy, which include wound care, pain medicine, and other standard instructions. The patient will be followed in the office with visits at 3 to 4weeks, and 3 months postoperatively.

At these visits, they will be assessed for postoperative complications including but not limited to: bleeding, urinary retention, fecal impaction, hospital re-admission and pain. Delayed complications -greater than four weeks- will be followed including impaired healing, constipation, abscess, fistula formation, fissure, and stenosis. The patient's pain score and type and amount of pain medications taken will be recorded by the patient daily for the first 2 weeks then weekly for a month postoperatively. This will be assessed using a pain diary which includes a visual analog pain scale (allowing the patient to describe their pain level on a scale between 1 and 10) and space to note the quantity of pain medications used. During each office visit, the operating surgeon will evaluate the patient.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between ages 18 through 80
* American Society of Anesthesiologists (ASA) level I, II and III
* External hemorrhoids must be present and deemed sufficiently symptomatic to warrant removal
* Internal hemorrhoids at least Grade II
* Must be able to be seen post-operatively by the surgeon at 3 to 4 weeks and 3 months after surgery

Exclusion Criteria:

* American Society of Anesthesiologists (ASA) level IV
* Grade I internal hemorrhoids
* Currently receiving coumadin, plavix, or other anticoagulants
* No prior sphincterotomy, drainage of abscess, fistulotomy, or similar procedures
* No pregnant women at the time of surgery
* No lactating women
* No inflammatory bowel disease
* No history of chronic, active hepatitis B, C, or HIV infection
* No prior chronic narcotic use (more than 30 days)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2011-08; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Post-operative complications | 3 to 4 weeks
  Patients will be assess for postoperative complications including but not limited to: bleeding, urinary retention, fecal impaction, hospital re-admission and pain.

SECONDARY OUTCOMES:
Delayed Post-Operative Complications | 3 months
  Delayed complications (greater than 4 weeks) will be followed including impaired healing, constipation, abscess, fistula formation, fissure, and stenosis.
Post-Operative Pain | 1 month
  The patient's pain score and type and amount of pain medications taken will be recorded by the patient daily for the first 2 weeks then weekly for a month postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Billingham, MD, Principal Investigator — Swedish Medical Center
Locations (1):
- Swedish Medical Center Colon Rectal Clinic, Seattle, Washington, United States